CLINICAL TRIAL: NCT03277326
Title: Randomised, Controlled Trial Comparing Interscalene Versus Anterior and Posterior Approaches of Suprascapular Nerve Block for Shoulder Arthroscopic Surgeries
Brief Title: Interscalene vs Anterior and Posterior Suprascapular Nerve Block for Shoulder Arthroscopic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/2459
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Arthroscopic Shoulder Surgery; Interscalene Block; Suprascapular Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ISB (Active Comparator): Interscalene brachial plexus block
  Interventions: Procedure: ISB
- aSSB (Active Comparator): Anterior Suprascapular Block
  Interventions: Procedure: aSSB
- pSSB (Active Comparator): Posterior Suprascapular Block
  Interventions: Procedure: pSSB

INTERVENTIONS:
Procedure: ISB — ISB block with 0.5% ropivicaine 15mls ( 45mg )
  Arms: ISB
Procedure: aSSB — aSSB block with 0.5% ropivicaine 15mls ( 45mg )
  Arms: aSSB
Procedure: pSSB — pSSB block with 0.5% ropivicaine 15mls ( 45mg )
  Arms: pSSB

SUMMARY:
To compare ISB vs anterior and posterior approaches of suprascapular block in terms of lung function and analgesia

DETAILED DESCRIPTION:
Interscalene block (ISB) is commonly used to provide pain control for shoulder surgeries. However, it is associated with several side effects, in particular, a high incidence of phrenic nerve blockade.

The suprascapular nerve block (SSB) has been proposed as an alternative to the ISB as it has a lower likelihood of causing phrenic nerve blockade. There are 2 commonly used approaches for the suprascapular nerve block, anterior and posterior. The anterior approach may still result in some degree of impairment of lung function.

The primary aim is to assess the pulmonary function after performance of ISB, aSSB and pSSB. Secondary outcomes are analgesic effects and incidence of adverse effects of these blocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective arthroscopic shoulder surgery under general anaesthesia
* Patients 21 years old and above
* American Society of Anesthesiologists (ASA) physical status 1 to 3
* BMI 18-35 kg/m2

Exclusion Criteria:

* Patients unable to give consent or inability to communicate/ cooperate
* Patients with chronic use of strong opioids (morphine, oxycodone)
* Patients with allergy to local anaesthetics or any drugs included in the study
* Patients with contraindications for regional anaesthesia such as coagulopathy
* Patients with pre-existing neurological deficits in upper limb/ phrenic nerve palsy
* Patients with pre-existing lung disease (COPD, uncontrolled asthma)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 2 years
  To assess the pulmonary function after performance of interscalene, anterior and posterior approaches to the suprascapular block

SECONDARY OUTCOMES:
Analgesic effects and complications | 2 years
  Analgesic effect (pain scores, opioid consumption, opioid related side effects), degree of motor blockade and incidence of adverse effects of blocks (Horner's syndrome, hoarseness of voice)

CONTACTS AND LOCATIONS:
Overall Officials: Yean Chin Lim, Principal Investigator — CGH
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No